CLINICAL TRIAL: NCT00659594
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Using the Environmental Exposure Chamber (EEC) to Assess the Onset of Action of Ciclesonide, Applied as a Nasal Spray (200 mg, Once Daily), in the Treatment of Seasonal Allergic Rhinitis (SAR) in Patients 18 Years and Older
Brief Title: Study Using the Environmental Exposure Chamber (EEC) to Assess the Onset of Action of Ciclesonide, Applied as a Nasal Spray in Treatment of Seasonal Allergic Rhinitis (BY9010/M1-406)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: BY9010/M1-406
Record Dates: First submitted 2008-04-14; First posted 2008-04-16 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-10

CONDITIONS: Rhinitis, Allergic, Seasonal; Hay Fever
Keywords: Seasonal Allergic rhinitis; Ciclesonide; Hay Fever; SAR
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — ciclesonide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator): Ciclesonide 200µg
  Interventions: Drug: Ciclesonide
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciclesonide — 200µg Ciclesonide versus Placebo
  Arms: 1
Drug: Placebo — placebo
  Arms: 2

SUMMARY:
The primary objective of this placebo-controlled EEC study is to determine the time to onset of action of ciclesonide, applied as a nasal spray (200 mg, once daily) in patients with SAR.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent signed and dated by the subject before conducting any study related procedure.
2. Male or female patients 18 years and older.
3. General good health, and free of any concomitant conditions or treatment that, in the judgment of the investigator, could interfere with study conduct, influence the interpretation of study observations/results, or put the patient at increased risk during the trial.
4. A history of SAR to short ragweed pollen for a minimum of two years immediately preceding the study entry. In the investigator's judgment, the SAR during this two- year period must have been of sufficient severity and would be expected to require treatment during the ragweed season.
5. A demonstrated sensitivity to short ragweed pollen known to induce SAR through a standard skin prick test. A positive test is defined as a wheal diameter of at least 3 mm larger than the diluent (negative) control wheal for the skin prick test. Documentation of a positive result 12 months prior to Screening Visit (B0) is acceptable.
6. Female is of child-bearing potential and is currently using and will continue to use a medically reliable method of contraception for the entire study duration (e.g. oral, injectable, trans-cutaneous or implantable contraceptives or intrauterine devices or double-barrier protection). Females who are not sexually active must agree to use double-barrier protection should they become sexually active during the course of the study. Women of child-bearing potential, or less than 1 year postmenopausal, will require a negative urine pregnancy test at the Screening Visit (B0) as well as prior to initiation of treatment at Treatment Visit (T0).Female subjects will be considered of non-childbearing potential and will not require a urine pregnancy test if at least one of the following apply:

   * Before menarche;
   * More than one year postmenopausal;
   * Had a hysterectomy;
   * Had a bilateral ovariectomy or salpingectomy or tubal ligation;
   * Have a congenital sterility.
7. Capable of understanding the requirements, risks, and benefits of study participation, and, as judged by the investigator, is capable of giving informed consent, will comply with all study requirements (visits, record keeping, etc), is suitable to participate, and will provide conscientious cooperation over the duration of the study and possesses the characteristics suitable to undertake this study.
8. Willingness to undergo a minimum of one (1) up to a maximum of five (5) priming sessions with short ragweed pollen in the EEC.

Exclusion Criteria:

1. Pregnancy, nursing, or plans to become pregnant or donate gametes (ova or sperm) for in vitro fertilization during the study period or for 30 days following the study period. Females unwilling to employ appropriate contraceptive measures to ensure that pregnancy will not occur during the study will be excluded.
2. Have clinically significant physical findings of nasal anatomical deformities causing greater than 50% obstruction based upon the clinical estimate by the investigator, including nasal polyps, septal defects or other clinically significant respiratory tract malformations, recent nasal biopsy, nasal trauma, or surgery and atrophic rhinitis or rhinitis medicamentosa (within the last 60 days prior to Screening Visit - B0).
3. Participation in any investigational drug trial within the 30 days preceding the Screening Visit (B0) and thereafter.
4. A known hypersensitivity to any corticosteroid or any of the excipients in the formulation.
5. History of severe respiratory infection or disorder [including, but not limited to bronchitis, pneumonia, chronic sinusitis, influenza, severe acute respiratory syndrome (SARS)] within the 14 days preceding the Screening Visit (B0).
6. History of alcohol or drug abuse within the preceding two years from Screening Visit (B0).
7. History of a positive test for HIV, hepatitis B or hepatitis C.
8. Active asthma requiring treatment with inhaled or systemic corticosteroids and/or routine use of b-agonists or any controller drugs (e.g. theophylline, leukotriene antagonist); intermittent use (less than or equal to 3 uses per week) of inhaled short-acting b-agonists is acceptable.
9. Use of any prohibited concomitant medications within the prescribed (per protocol) exclusion periods (refer to Section 6.3 of the protocol).
10. Use of antibiotic therapy for acute conditions within 14 days prior to the Screening Visit (B0) and thereafter. Low doses of antibiotics taken for prophylaxis are permitted if the therapy was started prior to the Screening Visit (B0) AND is expected to continue through out the Baseline Period (B0 to T0 Visit) and Treatment Visit (T0).
11. Initiation of immunotherapy during the study period or dose escalation during the study period. However, initiation of immunotherapy 90 days or more prior to the Screening Visit (B0) AND use of a stable (maintenance) dose (30 days or more prior to the Screening Visit (B0)) may be considered for inclusion provided no immunotherapy injections are received within 48 hours prior to a ragweed pollen exposure visit.
12. Previous participation in an intranasal ciclesonide study.
13. Non-vaccinated exposure to or active infection with, chickenpox or measles within the 21 days preceding the Screening Visit (B0).
14. Exposure to systemic corticosteroids for any indication, chronic or intermittent (e.g., arthritis), during the past 60 days from Screening Visit B0), or presence of an underlying condition that can reasonably be expected to require treatment with corticosteroids during the course of the study.
15. Use of topical corticosteroids in concentrations in excess of 1% hydrocortisone for dermatological conditions within 30 days prior to the Screening Visit (B0), or presence of an underlying condition that can reasonably be expected to require treatment with such preparations during the course of the study (B0 to T0 Visit, both visits inclusive). Hydrocortisone of less than or equal to 1% concentration covering less than or equal to 10% of the total body surface without occlusion is acceptable.
16. History of epilepsy or seizures (excluding febrile seizures).
17. History of coronary artery disease, uncontrolled hypertension, or other clinically significant cardiovascular disease.
18. Have any of the following conditions that are judged by the investigator to be clinically significant and/or affect the subject's ability to participate in the clinical trial:

    * Impaired hepatic function including alcohol related liver disease or cirrhosis;
    * Glaucoma;
    * Any systemic infection;
    * Hematological, renal, endocrine (except for controlled diabetes mellitus or postmenopausal symptoms or hypothyroidism);
    * Gastrointestinal disease;
    * Malignancy (excluding basal cell carcinoma);
    * A current neuropsychiatric condition with or without drug therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2004-11; Primary Completion 2005-02 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Time to onset of action, measured by a difference from placebo in the change from baseline in patient -assessed instantaneous TNSS following treatment | 14 hours

SECONDARY OUTCOMES:
Changes in TNSS from baseline at each time point | 14 hours
Changes in individual nasal symptom score from baseline at each time point | 14 hours
Proportion of patients exhibiting good/excellent response at each time point defined as all components of the patient-assessed TNSS scored as mild or less in severity | 14 hours
Spontaneous and elicited adverse events (AEs) | 14 hours
Physical exam (including nasal exam) | 14 hours
Vital signs | 14 hours

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (1):
- Altana/Nycomed, Mississauga, Ontario, Canada

REFERENCES:
- See also: BY9010-M1-406-RDS-2005-08-25.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4534&filename=BY9010-M1-406-RDS-2005-08-25.pdf